CLINICAL TRIAL: NCT00419458
Title: Respiratory Muscle Training in Ventilator Dependent Patients
Brief Title: Inspiratory Muscle Training in Ventilator Dependent Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NICHD 5R01HD42705
Record Dates: First submitted 2007-01-04; First posted 2007-01-08 (Estimated); Last update posted 2009-11-09 (Estimated); Status verified 2009-11

CONDITIONS: Failure to Wean; Respiratory Failure; Ventilator Dependent
Keywords: ventilator weaning; weaning; respiratory failure; inspiratory muscle strength training
MeSH Terms: conditions — Respiratory Insufficiency

INTERVENTIONS:
Procedure: inspiratory muscle strength training

SUMMARY:
The purpose of this study is to determine if inspiratory muscle strength training will increase the proportion of ventilator dependent patients weaned versus Sham treated patients.

DETAILED DESCRIPTION:
The inspiratory muscle strength training consists of 4 sets of 6-10 breaths through a threshold inspiratory muscle strength training device, 5 days per week. The inspiratory muscle training is conducted at the highest pressure setting tolerated by the patients. The Sham groups uses an inspiratory muscle trainer that does not increase inspiratory muscle strength. Both the treated and Sham groups participate in progressively lengthening periods of breathing without ventilator as tolerated. Patients are considered weaned when they can breathe for 72 consecutive hours without any ventilator support.

ELIGIBILITY:
Inclusion Criteria:

* Failure to wean patients in the medial, surgical and intermediate respiratory care units at Shands Hospital
* medically stable
* able to initiate spontaneous breaths
* able to provide informed consent
* able to follow simple instructions

Exclusion Criteria:

* life expectancy < 12 months due to malignancy
* damaged phrenic nerves
* neuromuscular diseases
* heart or lung transplant

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2004-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
ventilator dependent status

SECONDARY OUTCOMES:
breathing patterns during failed and passed unsupported breathing trials
maximal inspiratory pressure

CONTACTS AND LOCATIONS:
Overall Officials: Anatole D Martin, Ph D, PT, Principal Investigator — University of Florida; Andrea Gabrielli, MD, Study Director — University of Florida; Paul Davenport, Ph D, Study Director — University of Florida; Joseph Layon, MD, Study Director — University of Florida; Maher Baz, MD, Study Director — University of Florida; Lawrence Caruso, MD, Study Director — University of Florida; Ricardo Gonzalez-Rothi, MD, Study Director — University of Florida; Elosie Harman, MD, Study Director — University of Florida; Micheal Banner, Ph D, Study Director — University of Florida
Locations (1):
- Deprtment of Physical Therapy/Shands Hospital at the University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Ozcan MS, Bonett SW, Martin AD, Gabrielli A, Layon AJ, Banner MJ. Abnormally increased power of breathing as a complication of closed endotracheal suction catheter systems. Respir Care. 2006 Apr;51(4):423-5. No abstract available. PMID 16569266
- [Derived] Martin AD, Smith BK, Davenport PD, Harman E, Gonzalez-Rothi RJ, Baz M, Layon AJ, Banner MJ, Caruso LJ, Deoghare H, Huang TT, Gabrielli A. Inspiratory muscle strength training improves weaning outcome in failure to wean patients: a randomized trial. Crit Care. 2011;15(2):R84. doi: 10.1186/cc10081. Epub 2011 Mar 7. PMID 21385346